CLINICAL TRIAL: NCT03184402
Title: Efficacy and Safety of DWJ1252 in the Treatment of Functional Dyspepsia: A Multicenter, Randomized, Double-blind, Active-controlled Study (PART 2)
Brief Title: Efficacy and Safety of DWJ1252 in the Treatment of Functional Dyspepsia (PART 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DW_DWJ1252003
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Functional Dyspepsia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWJ1252 (Experimental)
  Interventions: Drug: DWJ1252; Drug: Placebo of Gasmotin
- Gasmotin (Active Comparator)
  Interventions: Drug: Gasmotin; Drug: Placebo of DWJ1252

INTERVENTIONS:
Drug: DWJ1252 — tablet
  Arms: DWJ1252
Drug: Gasmotin — tablet
  Arms: Gasmotin
Drug: Placebo of Gasmotin — tablet
  Arms: DWJ1252
Drug: Placebo of DWJ1252 — tablet
  Arms: Gasmotin

SUMMARY:
The purpose of this study is to evaluate the Efficacy and Safety of DWJ1252 in treatment of Functional Dyspepsia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female of at least 19 years old
* Patient with functional dyspepsia met the ROME III criteria

Exclusion Criteria:

* Patients with previous gastrointestinal surgery
* Patients with history of gastrointestinal bleeding, mechanical obstruction, perforation
* Patients with history of gastrointestinal cancer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
The change from baseline in GIS (Gastrointestinal Symptom Score) | At 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: SMG-SNU BORAMAE MEDICAL CENTER, Study Chair — SMG-SNU Boramae Medical Center
Locations (1):
- Smg-Snu Boramae Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No